CLINICAL TRIAL: NCT06186206
Title: Culturally and Linguistically Appropriate Vaccine Education (CLAVE): an Evaluation of Social Media Vaccine Communication Messages in Rural Guatemala
Brief Title: Culturally and Linguistically Appropriate Vaccine Education
Acronym: CLAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Stanford University (Other); Wuqu' Kawoq, Maya Health Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 00123120
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Vaccine Hesitancy
Keywords: Vaccination; Indigenous Communities; Social Media Campaign; Guatemala
MeSH Terms: conditions — Vaccination Hesitancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Social Media Messaging Only (Experimental): In this arm of the clinical trial, four selected communities will receive a culturally tailored social media campaign designed to increase childhood routine and HPV vaccine confidence and uptake. The campaign will be deployed via Facebook and will geographically target these communities. This arm serves as the first intervention group.
  Interventions: Behavioral: Social media interventions for vaccine uptake
- Social Media and Health Worker WhatsApp (Experimental): In this arm, another set of four communities will receive both the culturally tailored social media campaign (deployed via Facebook) and WhatsApp-based vaccine training for community healthcare workers. This arm serves as the second intervention group.
  Interventions: Behavioral: Social media interventions for vaccine uptake
- No Intervention (Control) (No Intervention)

INTERVENTIONS:
Behavioral: Social media interventions for vaccine uptake — Culturally Tailored Social Media Campaign: 4 communities receive a culturally tailored social media campaign via Facebook, focusing on geographical targeting. Content aligns with indigenous cultural norms and values, featuring educational materials, testimonials, and messaging addressing vaccine misconceptions on childhood routine and HPV vaccinations' importance and safety.
  WhatsApp-Based Vaccine Training for CHW: 4 communities receive both the culturally tailored social media campaign and WhatsApp-based vaccine training for CHWs. Interactive training allows CHWs to engage in discussions, seek guidance, and enhance their ability to communicate effectively. This component targets vaccine hesitancy and boosts vaccine uptake rates.
  Arms: Social Media Messaging Only; Social Media and Health Worker WhatsApp

SUMMARY:
The goal of this clinical trial is to test the effectiveness of culturally tailored social media campaigns and WhatsApp-based vaccine training for healthcare workers in increasing childhood routine and HPV vaccine confidence and uptake in mainly indigenous rural communities in Guatemala.

Main Research Questions:

* Does a culturally tailored social media campaign, deployed via Facebook and geographically targeting randomly assigned communities, increase childhood routine and HPV vaccine confidence and uptake in mainly indigenous rural communities in Guatemala?
* Does WhatsApp-based vaccine training for community healthcare workers increase vaccine uptake in these communities?

Participants in this study will be involved in the following tasks:

Community Healthcare Worker WhatsApp Training: Community healthcare workers will participate in WhatsApp training sessions to enhance their knowledge and skills related to vaccine education and communication.

Pre-Post Surveys: Surveys will be collected from individuals who are caretakers of children under 5 recruited from local health facilities. A total of 600 people will participate in the surveys (200 from each study arm and 200 pre-intervention). Surveys will be conducted in Spanish, K'iche', and Kaqchikel languages to compare vaccination uptake, hesitancy, and barriers/facilitators of vaccination.

Researchers will compare the groups receiving the social media campaign and WhatsApp training to those with no intervention to determine the effects on childhood routine and HPV vaccine confidence and uptake in indigenous rural communities in Guatemala.

DETAILED DESCRIPTION:
This clinical trial seeks to address the challenge of improving childhood routine and HPV vaccine confidence and uptake in mainly indigenous rural communities in Guatemala. The study is designed with three distinct study arms to assess the effectiveness of culturally tailored interventions. The interventions include a social media campaign delivered via Facebook, as well as WhatsApp-based vaccine training for community healthcare workers. The ultimate goal is to determine whether these interventions have a positive impact on vaccination rates and confidence in the target communities.

The clinical trial is organized into three arms. The first arm comprises four communities that will receive only the culturally tailored social media campaign, designed to increase childhood routine and HPV vaccine confidence and uptake. This campaign is specifically targeted at these communities through geographic targeting on Facebook. The second arm includes four communities that will receive both the social media campaign and WhatsApp-based vaccine training for community healthcare workers. Finally, the third arm, serving as the control group, consists of four communities where there will be no intervention.

The primary research questions guiding this clinical trial are as follows:

1. Does the culturally tailored social media campaign, deployed via Facebook and geographically targeting randomly assigned communities, increase childhood routine and HPV vaccine confidence and uptake in mainly indigenous rural communities in Guatemala?
2. Does WhatsApp-based vaccine training for community healthcare workers increase vaccine uptake in these communities?

In the second arm of the study, community healthcare workers will actively participate in WhatsApp training sessions. These sessions are designed to enhance their knowledge and communication skills related to vaccine education and advocacy. They will be encouraged to use the WhatsApp platform to engage in discussions, ask questions, and support one another in their efforts to effectively communicate the importance of childhood vaccinations with their patients.

Additionally, the clinical trial includes the collection of pre-post surveys from individuals who are caretakers of children under 5 years old. These individuals will be recruited from local health facilities, with a total of 600 participants across the three arms (200 from each intervention group and 200 from the pre-intervention phase). Surveys will be conducted in Spanish, K'iche', and Kaqchikel languages, allowing for a comprehensive assessment of vaccination uptake, hesitancy, and barriers/facilitators of vaccination.

To evaluate the effectiveness of the interventions, researchers will conduct a thorough analysis, comparing the three study arms. The analysis will involve several components:

* Comparing the first arm, which receives social media messaging only, to the control group to assess the impact of the social media campaign.
* Comparing the second arm, receiving both social media messaging and healthcare worker WhatsApp training, to the control group to determine the combined impact of these interventions.
* Lastly, comparing the two intervention groups to each other to identify any differences in effectiveness between the interventions.

Statistical methods, including regression analysis and interrupted time series analysis, will be employed to assess the impact of the interventions on the primary outcomes, which include childhood routine and HPV vaccine confidence and uptake.

In conclusion, this clinical trial represents a rigorous effort to address vaccination challenges in indigenous rural communities in Guatemala. By leveraging social media campaigns and healthcare worker training via WhatsApp, the study aims to improve vaccine confidence and uptake, ultimately contributing to better public health outcomes in these underserved populations.

ELIGIBILITY:
Inclusion Criteria:

* speaks a local language,
* live in the area,
* over age 18 and
* cares for a child 5 years or younger

Exclusion Criteria:

* Not an adult,
* not on social media

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Vaccination of children < 5 years | 6 months
  Health facility clinic data about vaccinations for key under 5 years of age vaccinations and HPV. We will measure overall coverage of routine childhood vaccines (defined as having completed all recommended vaccines by age), as well as coverage by individual vaccine type.
  Caregiver report of childhood vaccinations in the last 3 months, collected via in person survey (yes/no responses to questions about specific recent vaccines given the age of the child)
Hesitancy for vaccination | 2 months after intervention
  Caregiver report of childhood vaccination hesitancy, collected via in person survey. Collected using the Vaccine Hesitancy Scale, which has been validated in rural Guatemala for childhood vaccination

SECONDARY OUTCOMES:
Vaccine knowledge | 2 months after intervention
  Increase in knowledge of childhood and HPV vaccines

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Diamond-Smith, PhD, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- Maya Health Alliance | Wuqu' Kawoq, Tecpán Guatemala, Departamento de Chimaltenango, Guatemala

IPD SHARING:
Plan to Share IPD: No